CLINICAL TRIAL: NCT01376388
Title: A 52-week, Multi-centre, Open-label Study to Evaluate the Safety and Tolerability of GSK573719 125 mcg Once-daily in Combination With GW642444 25 mcg Once-daily Via Novel Dry Powder Inhaler (nDPI) in Japanese Subjects With Chronic Obstructive Pulmonary Disease.
Brief Title: Long-term Safety Study for GSK573719/GW642444 in Japanese
Acronym: DB2115362
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115362
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Pharmacogenetics; GSK573719/GW642444
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK573719/GW642444 (Experimental): 125/25mcg
  Interventions: Drug: GSK573719/GW642444 Inhalation Powder

INTERVENTIONS:
Drug: GSK573719/GW642444 Inhalation Powder — GSK573719/GW642444 inhalation powder inhaled orally once daily for 52 weeks.

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of GSK573719/GW642444 Inhalation Powder 125/25 mcg once-daily. The product will be delivered via the Novel Dry Powder Inhaler (nDPI) over 52 weeks to Japanese subjects with Chronic Obstructive Pulmonary Disease (COPD). This is a multi-centre, open-label study evaluating the safety of GSK573719/GW642444 Inhalation Powder 125/25 mcg. Treatment will be given once-daily in the morning. The target enrolment is approximately 120 subjects at approximately 20 study centres in Japan. The total duration of subject participation will be 54-55 weeks, consisting of a 7-14 day run-in period, 52-week treatment period and 1-week follow-up period. Subjects meeting all of the inclusion criteria and none of the exclusion criteria at screening visit (Visit 1) will enter 7-14 day run-in period. The run-in period is provided for completion of baseline safety evaluations and to obtain baseline measures of COPD status. At Visit 2, eligible subjects will start to take GSK573719/GW642444 125/25 mcg, and enter the treatment period. This treatment will be delivered via the Novel Dry Powder Inhaler (nDPI) once daily in the morning for 52 weeks. One nDPI will contain 30 doses of study medication. Subjects will be instructed to administer medication once daily in the morning for the duration of the 52-week treatment period. Each subject should be advised to adhere to this dosing regimen throughout the study. There will be a total of 8 study visits including at screening (Visit 1), initiation of treatment (Visit 2), and at 4weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks (Visit 3 through Visit 8, respectively). Follow-up (Visit 9) will be conducted by the phone contact approximately 1 week following the completion/withdrawal of treatment period. A subject will be considered to have completed the study upon completion of the last on-treatment visit (Visit 8). At the end of the treatment period, subjects will be prescribed appropriate COPD medication at the investigator's discretion.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and tolerability of GSK573719/GW642444 Inhalation Powder 125/25 mcg once-daily. The product will be delivered via the Novel Dry Powder Inhaler (nDPI) over 52 weeks to Japanese subjects with Chronic Obstructive Pulmonary Disease (COPD). This is a multi-centre, open-label study evaluating the safety of GSK573719/GW642444 Inhalation Powder 125/25 mcg. Treatment will be given once-daily in the morning. The target enrolment is approximately 120 subjects at approximately 20 study centres in Japan. The total duration of subject participation will be 54-55 weeks, consisting of a 7-14 day run-in period, 52-week treatment period and 1-week follow-up period. Subjects meeting all of the inclusion criteria and none of the exclusion criteria at screening visit (Visit 1) will enter 7-14 day run-in period. The run-in period is provided for completion of baseline safety evaluations and to obtain baseline measures of COPD status. Cardiovascular medical history/risk factors will be assessed at baseline. The following information will be collected from subjects receiving study medication and recorded in the eCRF: demography (including gender, ethnic origin and date of birth, height, weight), medical history (including duration of COPD and smoking history), COPD exacerbation assessment (documented history of ≥1 COPD exacerbation that required antibiotics/systemic corticosteroids or hospitalization in the past 12 months), concurrent medical conditions, and concomitant medication. At Visit 2, eligible subjects will start to take GSK573719/GW642444 125/25 mcg, and enter the treatment period. This treatment will be delivered via the Novel Dry Powder Inhaler (nDPI) once daily in the morning for 52 weeks. One nDPI will contain 30 doses of study medication. Subjects will be instructed to administer medication once daily in the morning for the duration of the 52-week treatment period. Each subject should be advised to adhere to this dosing regimen throughout the study. There will be a total of 8 study visits including at screening (Visit 1), initiation of treatment (Visit 2), and at 4weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks (Visit 3 through Visit 8, respectively). Follow-up (Visit 9) will be conducted by the phone contact approximately 1 week following the completion/withdrawal of treatment period. A subject will be considered to have completed the study upon completion of the last on-treatment visit (Visit 8). At the end of the treatment period, subjects will be prescribed appropriate COPD medication at the investigator's discretion. Primary endpoint is incidence and severity of adverse events. Secondary endpoints are clinical laboratory tests (hematology, clinical chemistry), change from baseline in vital signs (pulse rate and systolic and diastolic pressure), and 12-lead Electrocardiogram (ECG) assessments. And other endpoints are change from baseline in trough Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC), number of puffs of supplemental use of salbutamol, percentage of rescue-free days, percentage of symptom-free days, mean symptom scores, incidence of COPD exacerbations, and COPD device preference questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient.
* A signed and dated written informed consent prior to study participation.
* Japanese subjects 40 years of age or older at screening.
* Male or female subjects (female subjects who have child bearing potential has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods used consistently and correctly).
* Diagnosis of COPD.
* 10 pack-year or greater history of cigarette smoking.
* Post-bronchodilator FEV1/FVC of <0.7.
* Predicted FEV1 of <80%.

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* A current diagnosis of asthma.
* Respiratory disorders other than COPD.
* Clinically significant non-respiratory diseases or abnormalities that are not adequate controlled.
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD.
* A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition.
* Hospitalization for COPD or pneumonia within 12 weeks prior to screening.
* Subjects with lung volume reduction surgery within the 12 months prior to screening.
* Abnormal and clinically significant ECG findings at screening.
* Significantly abnormal finding from clinical chemistry or hematology, tests at screening.
* Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day.
* Regular use (prescribed every day, not for as-needed use) of short-acting bronchodilators via nebulized therapy.
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to screening.
* A know or suspected history of alcohol or drug abuse within 2 years prior to screening.
* Affiliation with the investigational site.
* Previous use of GSK573719, GW642444, the GSK573719/GW642444 combination or the Fluticasone Furoate/GW642444 combination.
* Use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115362 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 participants (par.) comprised the All Subjects Enrolled Population (ASEP; all par. with records in the study database). One par. in the ASEP was withdrawn due to a Good Clinical Practice violation and was thus withdrawn from the Intent-to-Treat Population (comprised of all participants who received at least one dose of study drug; n=130).
Pre-assignment Details: Following screening and a 2-week Run-in Period, during which participants were evaluated for Baseline safety and chronic obstructive pulmonary disease (COPD) status, eligible participants entered a 52-week Treatment Period, followed by a Follow-up Period.
Groups:
- UMEC/VI 125/25 µg: Participants received GSK573719/GW642444 (UMEC/VI) 125/25 micrograms (µg) inhalation powder via a dry powder inhaler (DPI) once daily (OD) in the morning for 52 weeks.
Period: Overall Study
Arm/Group | UMEC/VI 125/25 µg
Started | 130
Completed | 112
Not Completed | 18
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- UMEC/VI 125/25 µg: Participants received UMEC/VI 125/25 µg inhalation powder via a DPI OD in the morning for 52 weeks.
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (7.86)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 120
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE) Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs (occuring at a frequency threshold of >=5%) and SAEs.
Time Frame: 52 weeks
Population: Intent-to-Treat (ITT) Population: all participants who had received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Participants
  Any AE | 113
  Any SAE | 16

2. Primary Outcome: Number of Participants With AEs Classified by the Indicated Maximum Grade Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. AEs were classified according to intensity based upon the investigators' clinical judgment. The intensity was categorized as: mild (an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities); moderate (an event that is sufficiently discomforting to interfere with normal everyday activities); or severe (an event that prevents normal everyday activities).
Time Frame: 52 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Participants
  Mild | 83
  Moderate | 20
  Severe | 10

3. Secondary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, and Total Neutrophil Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of the indicated laboratory parameters at following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data at the indicated time points were analyzed. The number of participants assessed for each parameter is indicated by ''n=X" in the category title.
Measure: Mean (Standard Deviation); unit: Percentage of cells in blood
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Percentage of cells in blood
  Basophils, BL (Week -2), n=130 | 0.54 (0.340)
  Basophils, Week 12, n=127 | 0.58 (0.424)
  Basophils, Week 24, n=122 | 0.59 (0.386)
  Basophils, Week 52, n=112 | 0.60 (0.615)
  Basophils, WD Visit, n=10 | 0.35 (0.246)
  Basophils, Week 24/WD, n=129 | 0.58 (0.382)
  Basophils, Week 52/WD, n=122 | 0.58 (0.597)
  Eosinophils, BL (Week -2), n=130 | 3.90 (3.752)
  Eosinophils, Week 12, n=127 | 3.73 (3.178)
  Eosinophils, Week 24, n=122 | 4.07 (4.694)
  Eosinophils, Week 52, n=112 | 3.54 (2.936)
  Eosinophils, WD Visit, n=10 | 2.10 (1.662)
  Eosinophils, Week 24/WD, n=129 | 3.97 (4.593)
  Eosinophils, Week 52/WD, n=122 | 3.42 (2.876)
  Lymphocytes, BL (Week -2), n=130 | 29.07 (8.471)
  Lymphocytes, Week 12, n=127 | 28.48 (7.703)
  Lymphocytes, Week 24, n=122 | 28.40 (8.620)
  Lymphocytes, Week 52, n=112 | 28.71 (7.906)
  Lymphocytes, WD Visit, n=10 | 21.28 (8.110)
  Lymphocytes, Week 24/WD, n=129 | 28.12 (8.636)
  Lymphocytes, Week 52/WD, n=122 | 28.10 (8.150)
  Monocytes, BL (Week -2), n=130 | 6.15 (1.758)
  Monocytes, Week 12, n=127 | 6.33 (1.727)
  Monocytes, Week 24, n=122 | 6.27 (1.541)
  Monocytes, Week 52, n=112 | 6.20 (1.827)
  Monocytes, WD Visit, n=10 | 7.44 (1.290)
  Monocytes, Week 24/WD, n=129 | 6.32 (1.541)
  Monocytes, Week 52/WD, n=122 | 6.30 (1.818)
  Total Neutrophils, BL (Week -2), n=130 | 60.34 (9.047)
  Total Neutrophils, Week 12, n=127 | 60.88 (8.880)
  Total Neutrophils, Week 24, n=122 | 60.67 (9.595)
  Total Neutrophils, Week 52, n=112 | 60.96 (8.714)
  Total Neutrophils, WD Visit, n=10 | 68.83 (8.296)
  Total Neutrophils, Week 24/WD, n=129 | 61.01 (9.538)
  Total Neutrophils, Week 52/WD, n=122 | 61.60 (8.915)

4. Secondary Outcome: Eosinophil Values, Total Neutrophil Values, Platelet Count, and White Blood Cell (WBC) Count at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurment of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data at the indicated time points were analyzed. The number of participants assessed for each parameter is indicated by ''n=X'' in the category title.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter (GI/L)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
10^9 cells/Liter (GI/L)
  Eosinophils, BL (Week -2), n=130 | 0.245 (0.2324)
  Eosinophils, Week 12, n=127 | 0.225 (0.1815)
  Eosinophils, Week 24, n=122 | 0.260 (0.3243)
  Eosinophils, Week 52, n=112 | 0.219 (0.1992)
  Eosinophils, WD Visit, n=10 | 0.135 (0.1031)
  Eosinophils, Week 24/WD, n=129 | 0.254 (0.3171)
  Eosinophils, Week 52/WD, n=122 | 0.212 (0.1942)
  Total Neutrophils, BL (Week -2), n=130 | 3.874 (1.2587)
  Total Neutrophils, Week 12, n=127 | 3.798 (1.2169)
  Total Neutrophils, Week 24, n=122 | 3.946 (1.5517)
  Total Neutrophils, Week 52, n=112 | 3.899 (1.5434)
  Total Neutrophils, WD Visit, n=10 | 4.860 (2.0869)
  Total Neutrophils, Week 24/WD, n=129 | 3.953 (1.5326)
  Total Neutrophils, Week 52/WD, n=122 | 3.978 (1.6060)
  Platelet Count, BL (Week -2), n=130 | 234.3 (54.92)
  Platelet Count, Week 12, n=127 | 238.6 (56.35)
  Platelet Count, Week 24, n=122 | 239.3 (59.54)
  Platelet Count, Week 52, n=112 | 233.8 (58.63)
  Platelet Count, WD Visit, n=10 | 232.0 (84.03)
  Platelet Count, Week 24/WD, n=129 | 240.0 (60.02)
  Platelet Count, Week 52/WD, n=122 | 233.6 (60.65)
  WBC Count, BL (Week -2), n=130 | 6.38 (1.588)
  WBC Count, Week 12, n=127 | 6.18 (1.443)
  WBC Count, Week 24, n=122 | 6.39 (1.803)
  WBC Count, Week 52, n=112 | 6.30 (1.892)
  WBC Count, WD Visit, n=10 | 6.88 (2.203)
  WBC Count, Week 24/WD, n=129 | 6.37 (1.778)
  WBC Count, Week 52/WD, n=122 | 6.35 (1.916)

5. Secondary Outcome: Hemoglobin, Albumin, and Total Protein Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/Withdrawal (WD)
Description: Blood samples were collected for the measurement of hemoglobin, albumin, and total protein at the following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data at the indicated time points were analyzed. The number of participants assessed for each parameter is indicated by "n=X" in the category title.
Measure: Mean (Standard Deviation); unit: Grams/Liter (G/L)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Grams/Liter (G/L)
  Hemoglobin, BL (Week -2), n=130 | 145.1 (13.35)
  Hemoglobin, Week 12, n=127 | 148.2 (13.02)
  Hemoglobin, Week 24, n=122 | 148.1 (13.58)
  Hemoglobin, Week 52, n=112 | 148.2 (14.02)
  Hemoblobin, WD Visit, n=10 | 146.6 (12.82)
  Hemoglobin, Week 24/WD, n=129 | 148.0 (13.53)
  Hemoglobin, Week 52/WD, n=122 | 148.0 (13.88)
  Albumin, BL (Week -2), n=130 | 42.5 (2.58)
  Albumin, Week 12, n=127 | 42.9 (2.44)
  Albumin, Week 24, n=122 | 42.4 (2.76)
  Albumin, Week 52, n=112 | 41.9 (2.96)
  Albumin, WD Visit, n=10 | 41.3 (3.68)
  Albumin, Week 24/WD, n=129 | 42.3 (2.80)
  Albumin, Week 52/WD, n=122 | 41.9 (3.01)
  Total Protein, BL (Week -2), n=130 | 70.9 (4.20)
  Total Protein, Week 12, n=127 | 71.8 (4.50)
  Total Protein, Week 24, n=122 | 71.2 (4.20)
  Total Protein, Week 52, n=112 | 70.8 (4.78)
  Total Protein, WD Visit, n=10 | 68.7 (5.46)
  Total Protein, Week 24/WD, n=129 | 71.0 (4.22)
  Total Protein, Week 52/WD, n=122 | 70.6 (4.85)

6. Secondary Outcome: Hematocrit Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of hematocrit at the following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants remaining in the study and contributing evaluable data at the indicated time points were analyzed. The number of participants assessed at each time point is indicated by "n=X" in the category title.
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Proportion
  BL (Week -2), n=130 | 0.4460 (0.03857)
  Week 12, n=127 | 0.4534 (0.03575)
  Week 24, n=122 | 0.4515 (0.03720)
  Week 52, n=112 | 0.4517 (0.04063)
  WD Visit, n=10 | 0.4473 (0.03970)
  Week 24/WD, n=129 | 0.4512 (0.03724)
  Week 52/WD, n=122 | 0.4513 (0.04041)

7. Secondary Outcome: Alkaline Phosphatase (AP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatine Kinase, and Gamma Glutamyl Transferase (GGT) Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the WD Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
International Units/Liter (IU/L)
  AP, BL (Week -2), n=130 | 242.1 (80.70)
  AP, Week 12, n=127 | 250.2 (82.01)
  AP, Week 24, n=122 | 257.3 (81.40)
  AP, Week 52, n=112 | 247.5 (77.43)
  AP, WD Visit, n=10 | 227.7 (74.24)
  AP, Week 24/WD, n=129 | 254.2 (80.75)
  AP, Week 52/WD, n=122 | 245.9 (77.07)
  ALT, BL (Week -2), n=130 | 20.0 (10.42)
  ALT, Week 12, n=127 | 21.9 (13.19)
  ALT, Week 24, n=122 | 20.8 (13.06)
  ALT, Week 52, n=112 | 21.2 (12.09)
  ALT, WD Visit, n=10 | 31.7 (28.79)
  ALT, Week 24/WD, n=129 | 21.1 (13.56)
  ALT, Week 52/WD, n=122 | 22.0 (14.29)
  AST, BL (Week -2), n=130 | 23.4 (7.35)
  AST, Week 12, n=127 | 25.0 (8.90)
  AST, Week 24, n=122 | 23.9 (9.62)
  AST, Week 52, n=112 | 24.3 (8.94)
  AST, WD Visit, n=10 | 41.1 (42.05)
  AST, Week 24/WD, n=129 | 24.7 (14.48)
  AST, Week 52/WD, n=122 | 25.7 (15.04)
  Creatine Kinase, BL (Week -2), n=130 | 114.1 (59.56)
  Creatine Kinase, Week 12, n=127 | 120.3 (111.89)
  Creatine Kinase, Week 24, n=122 | 100.8 (42.60)
  Creatine Kinase, Week 52, n=112 | 111.3 (59.60)
  Creatine Kinase, WD Visit, n=10 | 387.5 (971.63)
  Creatine Kinase, Week 24/WD, n=129 | 124.0 (271.90)
  Creatine Kinase, Week 52/WD, n=122 | 134.0 (281.54)
  GGT, BL (Week -2), n=130 | 47.1 (54.80)
  GGT, Week 12, n=127 | 49.1 (57.91)
  GGT, Week 24, n=122 | 49.1 (63.21)
  GGT, Week 52, n=112 | 53.9 (78.30)
  GGT, WD Visit, n=10 | 46.3 (26.29)
  GGT, Week 24/WD Visit, n=129 | 49.2 (61.82)
  GGT, Week 52/WD Visit, n=122 | 53.3 (75.37)

8. Secondary Outcome: Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Creatinine, and Uric Acid Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, the WD Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measuremnt of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micromoles/Liter (µM/L)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Micromoles/Liter (µM/L)
  Direct Bilirubin, BL (Week -2), n=130 | 3.736 (1.7659)
  Direct Bilirubin, Week 12, n=127 | 3.514 (1.6731)
  Direct Bilirubin, Week 24, n=122 | 3.350 (1.4975)
  Direct Bilirubin, Week 52, n=112 | 3.680 (1.6426)
  Direct Bilirubin, WD Visit, n=10 | 3.249 (0.5407)
  Direct Bilirubin, Week 24/WD, n=129 | 3.340 (1.4632)
  Direct Bilirubin, Week 52/WD, n=122 | 3.644 (1.5846)
  Indirect Bilirubin, BL (Week -2), n=130 | 7.064 (2.8991)
  Indirect Bilirubin, Week 12, n=127 | 6.975 (2.7725)
  Indirect Bilirubin, Week 24, n=122 | 6.728 (2.5424)
  Indirect Bilirubin, Week 52, n=112 | 7.008 (2.9302)
  Indirect Bilirubin, WD Visit, n=10 | 5.985 (2.4517)
  Indirect Bilirubin, Week 24/WD, n=129 | 6.641 (2.5348)
  Indirect Bilirubin, Week 52/WD, n=122 | 6.924 (2.8987)
  Total Bilirubin, BL (Week -2), n=130 | 10.799 (4.3585)
  Total Bilirubin, Week 12, n=127 | 10.489 (4.1067)
  Total Bilirubin, Week 24, n=122 | 10.078 (3.6643)
  Total Bilirubin, Week 52, n=112 | 10.687 (4.2603)
  Total Bilirubin, WD Visit, n=10 | 9.234 (2.8156)
  Total Bilirubin, Week 24/WD, n=129 | 9.982 (3.6261)
  Total Bilirubin, Week 52/WD, n=122 | 10.568 (4.1714)
  Creatinine, BL (Week -2), n=130 | 74.3036 (19.60971)
  Creatinine, Week 12, n=127 | 74.3047 (19.32910)
  Creatinine, Week 24, n=122 | 73.2633 (18.90496)
  Creatinine, Week 52, n=112 | 75.6609 (18.69402)
  Creatinine, WD Visit, n=10 | 71.8692 (10.60022)
  Creatinine, Week 24/WD, n=129 | 73.2692 (18.55960)
  Creatinine, Week 52/WD, n=122 | 75.3501 (18.16682)
  Uric Acid, BL (Week -2), n=130 | 357.8408 (81.73895)
  Uric Acid, Week 12, n=127 | 353.2737 (81.17581)
  Uric Acid, Week 24, n=122 | 348.2993 (80.93244)
  Uric Acid, Week 52, n=112 | 353.2687 (89.55111)
  Uric Acid, WD Visit, n=10 | 343.7944 (87.40840)
  Uric Acid, Week 24/WD, n=129 | 349.1799 (80.95415)
  Uric Acid, Week 52, n=122 | 352.4921 (89.06027)

9. Secondary Outcome: Calcium, Chloride, Glucose, Carbon Dioxide/Bicarbonate (CO2/HCO3), Potassium, Sodium, Phosphorous Inorganic, and Urea/Blood Urea Nitrogen (Urea/BUN) Values at Baseline (BL; Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Description: as for outcome 7
Time Frame: BL (Screening visit: Week -2), Week 12, Week 24, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimoles/Liter (MMOL/L)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Millimoles/Liter (MMOL/L)
  Calcium, BL (Week -2), n=130 | 2.2954 (0.09315)
  Calcium, Week 12, n=127 | 2.2948 (0.09903)
  Calcium, Week 24, n=122 | 2.2837 (0.09096)
  Calcium, Week 52, n=112 | 2.2765 (0.09993)
  Calcium, WD Visit, n=10 | 2.2829 (0.15878)
  Calcium, Week 24/WD, n=129 | 2.2842 (0.09439)
  Calcium, Week 52/WD, n=122 | 2.2770 (0.10506)
  Chloride, BL (Week -2), n=130 | 103.7 (2.65)
  Chloride, Week 12, n=127 | 105.7 (2.51)
  Chloride, Week 24, n=122 | 105.7 (2.70)
  Chloride, Week 52, n=112 | 105.5 (2.93)
  Chloride, WD Visit, n=10 | 104.2 (3.65)
  Chloride, Week 24/WD, n=129 | 105.6 (2.79)
  Chloride, Week 52/WD, n=122 | 105.4 (3.00)
  Glucose, BL (Week -2), n=130 | 6.4447 (1.86640)
  Glucose, Week 12, n=127 | 6.3343 (1.63238)
  Glucose, Week 24, n=122 | 6.7313 (2.20449)
  Glucose, Week 52, n=112 | 6.6325 (1.81891)
  Glucose, WD Visit, n=10 | 6.5280 (1.52070)
  Glucose, Week 24/WD, n=129 | 6.7085 (2.15445)
  Glucose, Week 52/WD, n=122 | 6.6239 (1.79105)
  CO2/HCO3, BL (Week -2), n=130 | 25.7 (2.32)
  CO2/HCO3, Week 12, n=127 | 25.1 (2.29)
  CO2/HCO3, Week 24, n=122 | 24.1 (2.31)
  CO2/HCO3, Week 52, n=112 | 23.8 (2.18)
  CO2/HCO3, WD Visit, n=10 | 24.3 (3.50)
  CO2/HCO3, Week 24/WD, n=129 | 24.2 (2.41)
  CO2/HCO3, Week 52/WD, n=122 | 23.9 (2.30)
  Potassium, BL (Week -2), n=130 | 4.29 (0.380)
  Potassium, Week 12, n=127 | 4.34 (0.384)
  Potassium, Week 24, n=122 | 4.33 (0.374)
  Potassium, Week 52, n=112 | 4.31 (0.362)
  Potassium, WD Visit, n=10 | 4.42 (0.301)
  Potassium, Week 24/WD, n=129 | 4.33 (0.366)
  Potassium, Week 52/WD, n=122 | 4.32 (0.357)
  Sodium, BL (Week -2), n=130 | 141.4 (2.09)
  Sodium, Week 12, n=127 | 142.3 (1.95)
  Sodium, Week 24, n=122 | 142.3 (2.03)
  Sodium, Week 52, n=112 | 141.4 (2.26)
  Sodium, WD Visit, n=10 | 140.4 (3.72)
  Sodium, Week 24/WD, n=129 | 142.2 (2.21)
  Sodium, Week 52/WD, n=122 | 141.4 (2.41)
  Phosphorous Inorganic, BL (Week -2), n=130 | 0.9714 (0.15901)
  Phosphorous Inorganic, Week 12, n=127 | 1.0124 (0.16447)
  Phosphorous Inorganic, Week 24, n=122 | 0.9975 (0.16216)
  Phosphorous Inorganic, Week 52, n=112 | 0.9448 (0.16492)
  Phosphorous Inorganic, WD Visit, n=10 | 0.9913 (0.17558)
  Phosphorous Inorganic, Week 24/WD, n=129 | 0.9985 (0.16349)
  Urea/BUN, BL (Week -2), n=130 | 0.9486 (0.16555)
  Phosphorous Inorganic, Week 52/WD, n=122 | 5.2660 (1.52578)
  Urea/BUN, Week 12, n=127 | 5.4764 (1.80029)
  Urea/BUN, Week 24, n=122 | 5.4998 (1.50802)
  Urea/BUN, Week 52, n=112 | 5.4570 (1.66582)
  Urea/BUN, WD Visit, n=10 | 5.4335 (2.05521)
  Urea/BUN, Week 24/WD, n=129 | 5.4856 (1.52903)
  Urea/BUN, Week 52/WD, n=122 | 5.4551 (1.69111)

10. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Blood pressure measurements included systolic blood pressure (SBP) and diastolic blood pressure (DBP). Blood pressure was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from Baseline was calculated as the assessment value at the time of interest minus the Baseline value. The WD visit was conducted for participants who withdrew at any point during the study. The Week 24/WD visit was conducted for participants who completed the Week 24 visit or withdrew before Week 24. The Week 52/WD visit was conducted for participants who completed the Week 52 visit or withdrew before Week 52.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed (represented by "n=X" in the category title). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Millimeters of Mercury (mmHg)
  SBP, Week 4, n=128 | 1.1 (12.27)
  SBP, Week 8, n=127 | 2.0 (13.79)
  SBP, Week 12, n=127 | 2.5 (13.62)
  SBP, Week 24, n=122 | 2.7 (14.80)
  SBP, Week 36, n=116 | -3.3 (13.80)
  SBP, Week 52, n=112 | 0.4 (13.82)
  SBP, WD Visit, n=10 | -2.3 (18.62)
  SBP, Week 24/WD, n=129 | 2.5 (15.09)
  SBP, Week 52/WD, n=122 | 0.2 (14.19)
  DBP, Week 4, n=128 | 1.0 (9.21)
  DBP, Week 8, n=127 | 1.4 (9.99)
  DBP, Week 12, n=127 | 0.9 (10.71)
  DBP, Week 24, n=122 | 0.9 (10.81)
  DBP, Week 36, n=116 | -1.5 (11.10)
  DBP, Week 52, n=112 | 0.6 (10.23)
  DBP, WD Visit, n=10 | -2.0 (11.05)
  DBP, Week 24/WD, n=129 | 0.6 (10.92)
  DBP, Week 52/WD, n=122 | 0.4 (10.28)

11. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from Baseline was calculated as the assessment value at the time of interest minus the Baseline value. The WD visit was conducted for participants who withdrew at any point during the study. The Week 24/WD visit was conducted for participants who completed the Week 24 visit or withdrew before Week 24. The Week 52/WD visit was conducted for participants who completed the Week 52 visit or withdrew before Week 52.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: ITT Population. Only those participants with post-Baseline data available at the indicated time points were analyzed (represented by "n=X" in the category title). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Beats per minute
  Week 4, n=128 | -0.7 (10.21)
  Week 8, n=127 | -0.7 (9.39)
  Week 12, n=127 | -1.4 (10.81)
  Week 24, n=122 | -0.5 (10.63)
  Week 36, n=116 | -2.2 (10.56)
  Week 52, n=112 | -0.7 (10.63)
  WD Visit, n=10 | 9.0 (10.46)
  Week 24/WD, n=129 | -0.1 (10.67)
  Week 52/WD, n=122 | 0.1 (10.90)

12. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings at the Indicated Time Points
Description: A 12-lead ECG was recorded in a supine position after the participant was kept at rest in this position for at least 5 minutes. Data are presented as clinically significant (CS) or not clinically significant (NCS) abnormal findings. An abnormal and significant ECG finding includes the presence of a QT interval corrected for heart rate (QTc interval) >500 milliseconds (msec) or an uncorrected QT interval >600 msec, for participants with Bundle Branch Block QTc >530 msec based on an average QTc value of triplicate ECGs. The study investigator determined if the abnormal ECG finding was CS or NCS. The WD visit was conducted for participants who withdrew at any point during the study. The Week 24/WD and Week 52/WD visits were conducted for participants who completed the Week 24 visit or withdrew before Week 24 and completed the Week 52 visit or withdrew before Week 52, respectively. The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening visit).
Time Frame: Baseline (Screening visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | UMEC/VI 125/25 µg
Number analyzed (Participants) | 130
Participants
  BL (Week -2), Abnormal NCS, n=130 | 45
  BL (Week -2), Abnormal CS, n=130 | 2
  Week 12, Abnormal NCS, n=127 | 50
  Week 12, Abnormal CS, n=127 | 2
  Week 24, Abnormal NCS, n=122 | 43
  Week 24, Abnormal CS, n=122 | 3
  Week 36, Abnormal NCS, n=116 | 45
  Week 36, Abnormal CS, n=116 | 2
  Week 52, Abnormal NCS, n=112 | 47
  Week 52, Abnormal CS, n=112 | 2
  WD Visit, Abnormal NCS, n=9 | 4
  WD Visit, Abnormal CS, n=9 | 0
  Week 24/WD, Abnormal NCS, n=128 | 46
  Week 24/WD, Abnormal CS, n=128 | 3
  Week 52/WD, Abnormal NCS, n=121 | 51
  Week 52/WD, Abnormal CS, n=121 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 53 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who had received one dose of study drug.
Arm/Group | GSK573719/GW642444
Serious Adverse Events (participants affected / at risk) | 16/130
Other Adverse Events (participants affected / at risk) | 70/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK573719/GW642444 (N=130)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Dysphagia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Radicular cyst (Gastrointestinal disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cor pulmonale (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Sudden death (General disorders) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Cerebral infarction (Nervous system disorders) | 1
Mania (Psychiatric disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK573719/GW642444 (N=130)
Nasopharyngitis (Infections and infestations) | 49
Bronchitis (Infections and infestations) | 13
Pharyngitis (Infections and infestations) | 9
Constipation (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.